CLINICAL TRIAL: NCT00560248
Title: The BEACON Registry: Best Expert Agreement for Care of Occult MI Nationally
Brief Title: The BEACON Registry: Best Expert Agreement for Care of Occult Myocardial Infarction (MI) Nationally
Acronym: BEACON
Status: Terminated | Type: Observational
Why Stopped: Loss of funding
Sponsor: The Cleveland Clinic (Other)
Collaborators: Heartscape Technologies, Inc. (Industry); Novella Clinical (Other); PharmaVigilant (Unknown)
Responsible Party: W. Frank Peacock, MD, Cleveland Clinic
Other Study IDs: CCF2007-001; CCF2007-001
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Chest Pain
Keywords: Chest Pain; STEMI; UA/NSTEMI; ACS; Emergency Department
MeSH Terms: conditions — Chest Pain; ST Elevation Myocardial Infarction; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Patients presenting to the Emergency Department with chest pain suspected to be of cardiac origin.

SUMMARY:
The purpose of this registry is to assess and improve the process of care and health outcomes of patients presenting to the Emergency Department with chest pain suspected to be of cardiac origin. The study will identify which methods facilitate the diagnosis and risk stratification of ST elevation myocardial infarction (STEMI) or non STEMI, including patients with occult myocardial infarction (MI), and result in a shorter time to definitive diagnosis and treatment.

DETAILED DESCRIPTION:
The BEACON Registry is a multi-center data collection and follow-up registry. Participating Sites will collect information on patients presenting to the Emergency Department (ED) with chest pain. The purpose of the BEACON Registry is to evaluate the impact of new technologies, practice patterns and initiatives on patient time to diagnosis, patient time to treatment, patient survival and overall economics.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with chest pain suspected to be of cardiac origin.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 1897 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Time to definitive diagnosis of STEMI, UA/NSTEMI and non-cardiac chest pain; time to disposition decision will be used as an objective measure of time to definitive diagnosis | Index hospitalization

SECONDARY OUTCOMES:
Time to treatment, economic outcomes and survival outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William F. Peacock, MD, Principal Investigator — The Cleveland Clinic; Deepak L. Bhatt, MD, Principal Investigator — VA Boston Healthcare System; Venugopal Menon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States